CLINICAL TRIAL: NCT03795454
Title: Singing Kangaroos - Infant Care With Combined Auditory Intervention and Kangaroo Care
Brief Title: Can Singing Kangaroo Improve Outcome of Preterm Infants
Acronym: SingKang
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: Helsinki University Central Hospital (Other); Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Vineta Fellman, professor, University of Helsinki
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00003181SK
Record Dates: First submitted 2018-11-30; First posted 2019-01-07 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-06

CONDITIONS: Neurocognitive Dysfunction; Language Development
Keywords: Kangaroo care; MEG; AERP; preterm infant
MeSH Terms: conditions — Cognition Disorders; Premature Birth | interventions — Singing

STUDY DESIGN:
Intervention Model Description: In Helsinki, block randomization, one intervention at the time in the hospital. In Stockholm, both groups simultaneously cared in the hospital
Who Masked: Outcomes Assessor
Masking Description: Assessors do not know the intervention that took place before outcome assessed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Singing Kangaroo (Experimental): The parent is singing during the skin-to -skin sessions Musical therapeutist gives the instructions
  Interventions: Behavioral: Singing
- Silent Kangaroo (No Intervention): The parent is silent during the skin-to -skin sessions Musical therapeutist gives the instructions

INTERVENTIONS:
Behavioral: Singing — Infant-directed singing and singing of self-invented songs, especially songs emerging from the interaction with the infant, are especially encouraged. The families will receive audio material of children's songs, lullabies, and lyrics of the lullabies to support them if they feel unable to accomplish the task otherwise.
  Arms: Singing Kangaroo

SUMMARY:
To assess whether a musical intervention (maternal/paternal singing) during the skin-to-skin sessions (Kangaroo care) would improve the language development of the preterm infant. Infants will be randomized to singing or silence during the Kangaroo care from the age corresponding to 30th gestational week until term age (40 gestational weeks).

DETAILED DESCRIPTION:
The outcomes are:

a 2- (3-)year neurodevelopmental follow up

- Bayley Scales of Infant and Toddler Development, Third Edition (in Finnish in Finland and in Swedish in Sweden)

At the age corresponding to term (40 gestational weeks)

* Auditory event related potentials (AERPs) in electroencephalography (EEG), in Helsinki cohort
* Auditory event related magnetic fields in magnetoencephalgraphy (MEG) in Karolinska cohort
* Parental stress with The State Trait Anxiety Inventory (STAI)

ELIGIBILITY:
Inclusion Criteria:

* preterm infants at 30th gestational week capable of being in Kangaroo care

Exclusion Criteria:

* intensive care preventing Kangaroo care

Ages: 7 Days to 6 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2013-05-03 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
Auditory cortical responses | Age corresponding to term, ie 40 gestational weeks
  Auditory Event-Related Potentials (AERPs) at full-term age will be recorded with multi-feature paradigm (MFP), in which the mismatch negativity (MMN) to 5 speech-related auditory features can be recorded in a short time period.
Parental anxiety | 3 months age
  Parents' state anxiety is measured using the STAI (State-Trait Anxiety Inventory, Spielberger, 1983) with 20 self-descriptive statements once per week until the infant leaves the hospital and once in two weeks until the infant reaches the corrected age of 3 months,

SECONDARY OUTCOMES:
Neurocognitive development, language development | 2 year of age
  "Bayley III" :- Bayley Scales of Infant and Toddler Develoment, Third Edition (in Finnish in Finland and in Swedish in Sweden)
  - The following scales will be used: Cognitive, Language, Motor, Language scale includes Expressive Language and Receptive Language Motor scale includes Fine Motorics and Gross Motorics
  All scale ranges will be included (i.e., minimum and maximum scores) required to interpret any values. For example, if the *total* score is reported, the *total* range should be provided. If *subscale* scores are reported, the range for each *subscale* should be provided.

CONTACTS AND LOCATIONS:
Overall Officials: Kaija Mikkola, M.D. PhD, Principal Investigator — Helsinki University Central Hospital

IPD SHARING:
Plan to Share IPD: No
Depending on the AERP and MEG results there might be a need/wish to share individual anonymised data

REFERENCES:
- [Result] Partanen E, Martensson G, Hugoson P, Huotilainen M, Fellman V, Aden U. Auditory Processing of the Brain Is Enhanced by Parental Singing for Preterm Infants. Front Neurosci. 2022 Apr 4;16:772008. doi: 10.3389/fnins.2022.772008. eCollection 2022. PMID 35444514
- [Result] Kostilainen K, Partanen E, Mikkola K, Wikstrom V, Pakarinen S, Fellman V, Huotilainen M. Repeated Parental Singing During Kangaroo Care Improved Neural Processing of Speech Sound Changes in Preterm Infants at Term Age. Front Neurosci. 2021 Sep 3;15:686027. doi: 10.3389/fnins.2021.686027. eCollection 2021. PMID 34539329
- [Result] Kostilainen K, Hugoson P, Haavisto A, Partanen E, Mikkola K, Huotilainen M, Pakarinen S, Furmark C, Aden U, Fellman V. No impact of parental singing during the neonatal period on cognition in preterm-born children at 2-3 years. Acta Paediatr. 2023 Jul;112(7):1471-1477. doi: 10.1111/apa.16788. Epub 2023 Apr 25. PMID 37026177